CLINICAL TRIAL: NCT04463095
Title: Esophageal Mucosal Changes in Long Standing Achalasia Cardia and Reversibility After Per Oral Endoscopic Myotomy ( POEM )
Brief Title: Esophageal Mucosal Changes in Achalasia Cardia and Reversibility After Per Oral Endoscopic Myotomy - A Pilot Study
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Dr, Asian Institute of Gastroenterology, India
Other Study IDs: POEM EM
Record Dates: First submitted 2020-06-12; First posted 2020-07-09 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2020-07

CONDITIONS: Histopathology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PER ORAL ENDOSCOPY MYOTOMY (POEM) — Peroral endoscopic myotomy (POEM)combines thelong-term efficacy of a myotomy with the benefits of an endoscopic, minimally invasive procedure.Other therapeutic options include endoscopic balloon dilatation and surgical myotomy. Endoscopic balloon dilatation is still widely performed because of its relative non-invasiveness and simplicity, but it has a relatively lower success rate and often requires multiple treatment sessions. Surgical myotomy has been thought to be the curative therapeutic choice for symptomatic achalasia. However, it requires skin incisions and additional anti-reflux surgical intervention.Unlike surgical myotomy, POEM preserves the anatomical integrity of the LES and possibly minimizes postoperative reflux.

SUMMARY:
Esophageal mucosal changes in long standing achalasia cardia and reversibility after per oral endoscopic myotomy - A pilot study

Aims and Objectives:

* To study mucosal changes in patients with achalasia cardia
* To study potential malignant histopathological findings in long standing achalasia cardia
* To assess reversibility of mucosal changes after POEM
* To study co-relation of mucosal histopathology with predictors of sub-mucosal fibrosis
* To study muscle biopsy by light microscopy and electron microscopy for viral inclusions

Materials and Methods:

* Study Area - Patients of achalasia cardia undergoing POEM in Asian Institute of Gastroenterology.
* Study Design - Cross sectional study

Inclusion Criteria:

•All patients of achalasia cardia who will undergo POEM and an esophageal mucosal biopsy at 3 months of follow up

Exclusion Criteria:

* Patients of achalasia cardia not undergoing POEM or an esophageal mucosal biopsy at 3 months of follow up
* Upper gastro-intestinal surgically altered anatomy ( apart from previous Heller Myotomy )
* Pregnancy
* Patients not giving consent for participation
* End Point( Length of follow up )- 3 months after POEM - single follow up.

Study Procedure:

Before POEM, all patients will undergo symptom evaluation, esophagogastroduodenoscopy (EGD), high resolution esophageal manometry and timed barium esophagogram.The diagnosis of achalasia will be based on a combination of clinical presentation, esophagogastroduodenoscopy, barium esophagogram and high resolution manometric findings.

Symptoms will be classified by using the Eckardt score.Type of Achalasia will be classified according to the Chicago classification. Esophagus shape (sigmoid vs nonsigmoid), presence of hiatus hernia, presence of esophagitis will be assessed on esophagogastroduodenoscopy. Duration since first symptoms of achalasia will be recorded.

All patients fulfilling the inclusion criteria will undergo Per Oral Endoscopic Myotomy (POEM). During POEM, a mucosal biopsy and a muscle biopsy of the Esophagus will be taken. Patients will be followed up at a single time, 3 months after POEM. During the follow up visit, patients will undergo esophagogastroduodenoscopy guided mucosal biopsy of the Esophagus. Patients will be divided into two groups based on the duration of symptoms of achalasia- Those having symptoms for 1 year or less and those having symptoms for more than 5 years. Histopathological changes in the Esophagus and reversibility of these changes after POEM will be compared between the two study groups to draw a conclusion.

DETAILED DESCRIPTION:
Introduction and Background:

Achalasia cardiais a rare, chronic, esophageal motility disorder with an estimated annual prevalence of 1 per 1,00,000 subjects. The disease can occur at all ages, but the incidence seems to increase with age. The predominant symptoms are dysphagia and regurgitation, because of the impaired relaxation of the lower esophageal sphincter (LES) and the loss of normal peristalsis.Achalasia is a neurodegenerative disease resulting from an inflammatory and/or autoimmune process ultimately leading to aganglionosis. The etiology and pathogenesis of achalasia is still unknown. The primary pathophysiologic abnormality is a loss of the intrinsic inhibitory innervation of the lower esophageal sphincter (LES) and the segment of smooth musculature of the esophageal body. The resultant denervation and reduction of post-ganglionic nerve fibers have been postulated to be related to the hypertensive or non-relaxing LES in patients with achalasia.Esophagectomy or surgical myotomy specimens have demonstratedabsence or reduction in ganglion cells as well as varying degrees of cytotoxic T-cell inflammation in the myenteric plexus of patients with achalasia. Studies demonstrating an association between achalasia and certain HLA phenotypes, and an increased immunologic response to Herpes Simplex Virus-1 (HSV-1) in the serum and LES myenteric plexusof achalasia patients further support the notion of inflammation playing a central role in pathogenesis.However, it is not known whether this inflammation is part of the process that leads to the loss of the plexus, or whether it is secondary to the outflow obstruction with consecutive stasis in achalasia. Persistent esophageal distension with retention of foods and fluids, bacterial overgrowth, and impaired clearance of regurgitated acid and gastric contents lead to chronic inflammation and passively cause dysplasia and carcinoma. The prognosis of patients who develop such carcinomas remains poor. The aim of therapy is to reduce food stasis, which might interrupt the progression to carcinoma and thus reduce the risk of squamous cell carcinoma.

No currently available treatment options result in regeneration of myenteric neurons to bring back esophageal motility. However, lowering LES pressure can significantly reduce symptoms and improve quality of life. To achieve this outcome (LES pressure reduction), therapeutic techniques have been modified from time to time. Graded pneumatic balloon dilatation (PBD) has replaced conventional one-time dilatation and open Heller's myotomy has cleared the way for laparoscopic Heller's myotomy (LHM) with fundoplication.Recently, per oral endoscopic myotomy (POEM) was introduced by Inoue et al. as a less invasive and effective curative treatment option with minimal complications.Peroral endoscopic myotomy (POEM)combines thelong-term efficacy of a myotomy with the benefits of an endoscopic, minimally invasive procedure.Other therapeutic options include endoscopic balloon dilatation and surgical myotomy. Endoscopic balloon dilatation is still widely performed because of its relative non-invasiveness and simplicity, but it has a relatively lower success rate and often requires multiple treatment sessions. Surgical myotomy has been thought to be the curative therapeutic choice for symptomatic achalasia. However, it requires skin incisions and additional anti-reflux surgical intervention.Unlike surgical myotomy, POEM preserves the anatomical integrity of the LES and possibly minimizes postoperative reflux.

Rationale of the study:

* There have been very few studies systematically analysing the histopathological changes in the mucosa and muscle of the Esophagus in Achalasia Cardia.
* Therefore we want to study the histopathological changes in the mucosa and muscle of the Esophagus in achalasia cardia patients and observe how the histopathological changes differ between early achalasia cardia and long-standing achalasia cardia.
* Achalasia Cardia is a potential pre-malignant condition which can lead to esophageal carcinoma.
* Principal investogator want to study the pre-malignant and malignant changes in the Esophagus in achalasia cardia patients.
* Also want to study whether per oral endoscopic myotomy ( POEM ) reverses the histopathological and pre-malignant changes in the Esophagus.

ELIGIBILITY:
Inclusion Criteria:

* • All patients of achalasia cardia who will undergo POEM and an esophageal mucosal biopsy at 3 months of follow up

Exclusion Criteria:

* • Patients of achalasia cardia not undergoing POEM or an esophageal mucosal biopsy at 3 months of follow up

  * Upper gastro-intestinal surgically altered anatomy ( apart from previous Heller Myotomy )
  * Pregnancy
  * Patients not giving consent for participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Since the present study is pilot based in assessing the primary outcome, it has been decided to cover 30 patients and follow up at 3 months. Hence no power calculation is used to estimate the sample size.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
1.To study mucosal changes in patients with achalasia cardia | 12 weeks
  Number of ganglion cells will be measured in the mucosal biopsy (normal number of ganglion cells are 2 to 12 per mm on Histopathological examination). The size of the ganglion cells will be measured.(normal size of ganglion cells is 10 to 40 microns). Median number of neurons will be measured.(normal median number of neurons are 2 to 6 on histopathological examination).
2. To study potential malignant histopathological findings in long standing achalasia cardia | 12 weeks
  The mean Ki-67 and mean p53 positive ratio will be measured in the histopathological examination.

SECONDARY OUTCOMES:
3.To study co-relation of mucosal histopathology with predictors of sub-mucosal fibrosis | 12 weeks
  The fibrosis score will be measured in the histopathological examination.
4. To evaluate reversibility of mucosal changes after per oral endoscopic myotomy (POEM ) | 12 weeks
  Number of ganglion cells will be measured in the mucosal biopsy (normal number of ganglion cells are 2 to 12 per mm on Histopathological examination). The size of the ganglion cells will be measured.(normal size of ganglion cells is 10 to 40 microns). Median number of neurons will be measured.(normal median number of neurons are 2 to 6 on histopathological examination). These findings will be measured 12 weeks post POEM.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pranav Milind Ambardekar, MBBS MD, Principal Investigator — Asian institute of Gastroenterology/AIG Hospitals
Locations (1):
- Asian institute of Gastroenterology/AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No